CLINICAL TRIAL: NCT06521970
Title: Comparison of Dynamic Posture and Head Position in Kyphotic Individuals According to Gender
Brief Title: Dynamic Posture and Head Position in Kyphotic Female and Male
Acronym: DPHP
Status: Completed | Type: Observational
Sponsor: Gaziantep Islam Science and Technology University (Other)
Responsible Party: Principal Investigator, Gönül Elpeze, Assistant Proffessor, Gaziantep Islam Science and Technology University
Other Study IDs: GIBSTU
Record Dates: First submitted 2024-07-09; First posted 2024-07-26 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Kyphosis Thoracic; Postural, Thoracic Kyphosis; Postural Kyphosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Female: Thoracic kyphosis (TK) angle of ≥ 50° The kyphosis angle, dynamic postural performance, forward head position
  Interventions: Diagnostic Test: The kyphosis angle; Diagnostic Test: dynamic postural performance; Diagnostic Test: forward head position
- Male: Thoracic kyphosis (TK) angle of ≥ 50° The kyphosis angle, dynamic postural performance, forward head position
  Interventions: Diagnostic Test: The kyphosis angle; Diagnostic Test: dynamic postural performance; Diagnostic Test: forward head position

INTERVENTIONS:
Diagnostic Test: The kyphosis angle — The subject was positioned in a neutral standing position. the short side of the phone was placed on the T1-3 spinous process and the protractor was set to 0°. Subsequently, the phone was placed on the T12, and the angular value displayed on the screen was recorded as the kyphotic angle.
  Other Names: Thorasic kyphosis
Diagnostic Test: dynamic postural performance — The test measures spinal alignment deviations during static loading in the 90° shoulder flexion position. The test measurements are made in a standing position with arms 90° flexed, without weight, and after 30 seconds with weight.
  Other Names: Matthias Test
Diagnostic Test: forward head position — The individual stands with his heels and pelvis in contact with the wall. The severity of kyphosis is interpreted by measuring the distance between the occiput and the wall in cm with the head facing forward. The intensity of kyphosis is classified as mild (≤5 cm), moderate (5.1-8 cm) and severe (>8 cm)
  Other Names: Occiput-Wall Distance

SUMMARY:
This study examined the comparison of dynamic posture and head position in kyphotic ındividuals according to gender.

Methods: A total of 54 female and male adolescents (between the ages of 12 and 18) with a thoracic kyphosis (TK) angle of ≥ 50° were divided into two groups according to gender.

The kyphosis angle, dynamic postural performance, and forward head position were measured using a flexible ruler, Mathiass test, and occiput wall distance.

DETAILED DESCRIPTION:
This study examined the comparison of dynamic posture and head position in kyphotic ındividuals according to gender.

Methods: This observational cross-sectional study was conducted with 54 subjects. Subjects aged 12 to 18 years with a kyphosis angle of ≥50º and the children and their parents who agreed to participate in the study were included. Individuals with Scheurmann kyphosis, scoliosis (Cobb angle >10°), and other congenital spine abnormalities were excluded.

The kyphosis angle was measured using a smartphone inclinometer. Dynamic posture was assessed using the Matthias test. Head position was obtained using occiput-wall distance.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a kyphosis angle of ≥50º and the children and their parents who agreed to participate in the study were included.

Exclusion Criteria:

* Individuals with Scheurmann kyphosis, scoliosis (Cobb angle >10°), and other congenital spine abnormalities were excluded.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Study Population: ADOLESCENT
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2023-06-16 (Actual); Primary Completion 2024-01-20 (Actual); Study Completion 2024-06-05 (Actual)

PRIMARY OUTCOMES:
Matthias test | 1 year
  Matthias test assesses dynamic postural performance

SECONDARY OUTCOMES:
Occiput wall distance | 1 year
  Occiput wall distance is an assessment method to determine forward head posture in clinical settings.

CONTACTS AND LOCATIONS:
Overall Officials: Gonul Elpeze, Asst. Prof., Principal Investigator — Gaziantep Islam Science and Technology University Physical Therapy and Rehabilitation Department
Locations (1):
- Gaziantep Islam Science and Technology University, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No